CLINICAL TRIAL: NCT07152990
Title: Prevalence of Nocturnal Hypoventilation Diagnosed by Transcutaneous Oxy-capnography in a Population of Obese Subjects Fitted With Continuous Positive Airway Pressure for Obstructive Sleep Apnea Hypopnea Syndrome.
Brief Title: Prevalence of Nocturnal Hypoventilation in Obese Subjects Fiited With Continuous Positive Airway Pressure for Obstructive Sleep Apnea / Hypopnea Syndrome
Acronym: CAPNOSOH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fonds de dotation Agir pour les Maladies Chroniques (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/24/0290; 2025-A00694-45 (Other: ANSM)
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Nocturnal Hypoventilation; Obesity; Sleep Apnea Hypopnea Syndrome
Keywords: Nocturnal hypoventilation; obesity; sleep apnea syndrome; continuous positive pressure; transcutaneous capnography
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: All patients will undergo transcutaneous oxy-capnography and answer quality of life questionnaires. Only patients presenting nocturnal hypoventilation defined with PTcCO2 > 49 mmHg more than 10% of the time of capnographic recording will continue the study with additional interventions. Patients without nocturnal hypoventilation will finish the study after the capnographic recording visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese Patients with Obstructive Sleep Apnea/Hypopnea (Other)
  Interventions: Other: Transcutaneous Oxy-Capnography; Other: Quality of life questionnaires; Other: Arterial gasometry; Other: Body plethysmography; Other: Spirometry with reversibility test; Other: Clinical examination

INTERVENTIONS:
Other: Transcutaneous Oxy-Capnography — Patients will be monitored using transcutaneous oxy-capnography to evaluate the prevalence of nocturnal alveolar hypoventilation in these population. Nocturnal alveolar hypoventilation is defined with PTcCO2 > 49 mmHg more than 10% of the time of capnographic recording.
Other: Quality of life questionnaires — Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index, and the "Patient-Reported Hypoventilation Questionnaire".
Other: Arterial gasometry — Arterial blood gas analysis will be performed only in patients presenting nocturnal hypoventilation.
Other: Body plethysmography — Plethysmography will be performed only in patients presenting nocturnal hypoventilation. It will be used to measure lung volume and assess pulmonary function. This non-invasive procedure involves the patient breathing into a device that measures changes in pressure within a sealed chamber.
Other: Spirometry with reversibility test — The intervention will be performed only in patients presenting nocturnal hypoventilation. Spirometry with a reversibility test will be performed to assess lung function and evaluate the response to bronchodilators. The procedure involves measuring forced expiratory volume and forced vital capacity before and after the administration of a bronchodilator.
Other: Clinical examination — Clinical exam will be performed only in patients presenting nocturnal hypoventilation. It will consists of standard interview/clinical examination: vital signs, cardiological, pulmonary, abdominal, neurological examination, search for clinical signs of nocturnal hypoventilation, search for signs of hypoxia/hypercapnia, pulmonary auscultation.

SUMMARY:
CAPNOSOH study is a single-center study conducted at Toulouse University Hospital, aiming to estimate the prevalence of obese and apneic subjects maintaining nocturnal hypoventilation under continuous positive airway pressure (CPAP).

DETAILED DESCRIPTION:
Obstructive sleep apnea hypopnea syndrome (OSAS) is highly prevalent in the global population (1 in 10 people worldwide according to Inserm), particularly in relation to the increase in the prevalence of obesity. The standard treatment for this pathology is continuous positive airway pressure (CPAP) which most often allows, when properly applied and adjusted, the normalization of symptoms and the apnea-hypopnea index (AHI). In addition to OSAHS, some obese subjects are at risk of presenting hypoventilation obesity syndrome (OHS) defined by the presence of obesity (body mass index [BMI] > 30 kg/m2) associated with diurnal hypoventilation. (PaCO2 > 45 mmHg) in the absence of other respiratory pathology. Identifying patients with OS is often difficult but essential, as early as possible.

Transcutaneous capnography, when properly performed and interpreted, is a much more informative tool than nocturnal oximetry, and could therefore allow better screening for these patients. It is an examination increasingly used in pulmonology departments/sleep centers.

The CAPNOSOH study is a single-center study conducted at Toulouse University Hospital, aiming to estimate the prevalence of obese and apneic subjects maintaining nocturnal hypoventilation under continuous positive airway pressure (CPAP). The study hypothesis is based on the limited data present in the literature. This is preliminary work for a multicenter study aimed at determining the impact of nocturnal hypoventilation without daytime hypercapnia on the quality of life and morbidity and mortality of patients.

We estimate that between 10 to 20% of obese subjects on CPAP hypoventilate at night.

ELIGIBILITY:
Inclusion criteria:

* Obese patients (Body Mass Index > 30 kg/m2)
* Fitted by one of the following providers: ASTEN, Vitalaire, Orkyn, ISIS, RespiO2, BASTIDE for > 3 months with compliance of more than 4 consecutive hours per night in average during 3 months
* "Good quality" criteria for continuous positive airway pressure (CPAP) treatment: compliance > 4 consecutive hours per night, unintentional leaks < limit defined by the manufacturer, residual AHI < 10/h
* Aged 18 to 80
* Affiliated or beneficiaries of the social security system or equivalent
* Having given written informed consent
* Able to understand instructions and information given

Exclusion criteria :

* Patient under legal protection measure
* Non-compliant patients
* Pregnant or breast-feeding women (assessed on questioning)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Prevalence of nocturnal alveolar hypoventilation | 1 month
  Prevalence of nocturnal alveolar hypoventilation will be diagnosed by transcutaneous oxy-capnography. Nocturnal alveolar hypoventilation is defined with PTcCO2 > 49 mmHg more than 10% of the time of capnographic recording.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Toulouse Hôpital Larrey, Toulouse, Occitanie, France